CLINICAL TRIAL: NCT04272047
Title: Prevention of Lower Limb and Groin Injuries: the Sport Without Injury ProgrammE (SWIPE) Football Trial
Acronym: SWIPEsoccer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: The Swedish Research Council (Other Government); Swedish Research Council for Sport Science (Other)
Responsible Party: Principal Investigator, Martin Hägglund, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-06462
Record Dates: First submitted 2020-02-10; First posted 2020-02-17 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Athletic Injuries
Keywords: Prevention
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Intervention Model Description: This is a three-armed intervention study that evaluates the injury preventive effects of three different training interventions in youth and adult football players. Two intervention arms are randomized and one arm acts as a non-randomized comparison group.
Who Masked: Outcomes Assessor
Masking Description: Physiotherapists who assess injuries are blinded to group belonging. Statistician performing outcome analyses are blinded to group belonging.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Knee Control+ (Experimental): Knee Control+ consists of 6 different exercises, with 10 different variations/progressions, and takes 10-15 minutes to complete. In addition, teams are instructed to perform a 5-minute running warm-up before the Knee Control+ exercises. Teams are to carry out the running warm-up and Knee Control+ at all training sessions, and the running warm-up before all matches, during the whole season. Knee Control+ is based on the Knee Control program but with more variations for each exercise making it easier to tailor for the needs in the respective teams.
  Interventions: Other: Knee Control+ program
- Adductor strengthening program (Experimental): The Adductor strengthening program consists of a single exercise with three levels of difficulty. The exercise is based on the Copenhagen Adduction exercise. Teams are to carry out the Adductor strengthening program as part of their regular warm-up 2-3 times per week, one set per side, during the pre-season, and 1 time per week, one set per side during the in-season.
  Interventions: Other: Adductor strengthening program
- Knee Control (Active Comparator): Teams will carry on their normal training and warm-up routines using the Knee Control program with no intervention from the researchers. Knee Control consists of 6 different exercises, with 4 different variations/progressions and 1 pair-exercise.
  Interventions: Other: Knee Control program

INTERVENTIONS:
Other: Knee Control+ program — 15-20 minute training program to be performed at all team training sessions during the season.
  Arms: Knee Control+
Other: Adductor strengthening program — Adductor strengthening program to be performed 2-3 times per week, one set per side, during the pre-season, and 1 time per week, one set per side during the in-season.
  Arms: Adductor strengthening program
Other: Knee Control program — 15-20 minute training program to be performed as per the team's usual routines (no intervention from the researchers).
  Arms: Knee Control

SUMMARY:
This is a three-armed intervention study that evaluates the injury preventive effects of three different training interventions in youth and adult football players. Two intervention arms are randomized and one arm acts as a non-randomized comparison group. Half of randomized participants will receive a general injury prevention exercise program with emphasis on the lower extremities, and the other half a hip/groin focused injury prevention exercise. A third group of participants who already use an injury prevention exercise program at study inclusion are invited to participate as a non-randomized comparison group and continue their usual training practices.

DETAILED DESCRIPTION:
The study is a cluster-randomized controlled trial including male and female youth and adult football players (≥14 years). Club is used as cluster unit, where all the teams from the same club will be randomized to the same intervention arm. The randomization is stratified by level (junior/senior) and sex (male/female).

The study has three intervention arms:

Teams in the randomized intervention group A receive education of the injury prevention exercise program Knee Control+ (Knäkontroll+) before the start of the competitive football season in April. Knee Control+ consists of 6 different exercises, with 10 different variations/progressions, and takes 10-15 minutes to complete. In addition, teams are instructed to perform a structured 5-minute running warm-up before the Knee Control+ exercises. Teams are to carry out the running warm-up and Knee Control+ at all training sessions, and the running warm-up before all matches, during the whole season.

Teams in the randomized intervention group B receive education of an Adductor strengthening program before the start of the competitive football season in April. The Adductor strengthening program consists of a single exercise with three levels of difficulty, as described by Harøy et al., 2019, British Journal of Sports Medicine. The exercise is based on the Copenhagen Adduction exercise. Teams are to carry out the Adductor strengthening program as part of their regular warm-up 2-3 times per week, one set per side, during the pre-season, and 1 time per week, one set per side during the in-season. One set takes about 5 minutes to complete for a pair of players.

Teams reporting that they are already using the injury prevention exercise program Knee Control (Knäkontroll) at recruitment are not eligible for inclusion in the randomization. They will be invited to participate in the study as a non-randomized intervention group C and act as a comparison group to the randomized groups A and B. These teams will carry on their normal training and warm-up routines with no intervention from the researchers. Knee Control consists of 6 different exercises, with 4 different variations/progressions and 1 pair-exercise.

Hypotheses:

Hypothesis 1: Teams/athletes in the randomized group A (Knee Control+) will have a lower rate of ankle, knee and hamstring injuries compared to teams/athletes in the randomized group B (Adductor strengthening program).

Hypothesis 2: Teams/athletes in the randomized group B (Adductor strengthening program) will have a lower rate of hip/groin injuries compared to teams/athletes in the randomized group A (Knee Control+).

Hypothesis 3: Teams/athletes in the randomized group A (Knee Control+) will have a higher intervention compliance compared to teams/athletes in the non-randomized comparison group (Knee Control).

Data collection:

Teams are followed for one competitive football season from April to October 2020. Data registered for the study include individual exposure to football training and matches, and injuries that occur as a result of participation in football. Exposure and injury data are athlete-reported prospectively every week using web-based questionnaires (the Oslo Sports Trauma Research Center questionnaire). Study designated physiotherapists will collect additional injury information for the four main injury outcomes via telephone interview using a standard injury card. Use of the intervention (compliance) is reported weekly by the team coach and the athletes. Coaches and players will report demographics at baseline, and at three time-points during the season (baseline, mid-season, end of season) will report use and experiences of the training interventions, injury risk perceptions and outcome expectancies.

Sample size for primary outcomes:

Hypothesis 1: required sample size for primary outcome "any football related injury occurring to the ankle, knee or hamstrings, regardless of need of care or absence from football training or matches" is 252 subjects (approximately 17 teams). To account for a 30% dropout a sample size of 328 subjects (approximately 22 teams) is planned at study start.

Hypothesis 2: required sample size for primary outcome "any football related injury occurring to the hip/groin, regardless of need of care or absence from football training or matches" is 301 subjects (approximately 20 teams). To account for a 30% dropout a sample size of 391 subjects (approximately 26 teams) is planned at study start.

Statistical analysis plan:

Generalised estimating equations will be used to analyse cluster-aggregated weekly data of injuries and exposure. A Poisson distribution with a log link function will be applied to calculate the rate ratio and corresponding 95% confidence intervals for the injury incidence and injury prevalence according to the intention to treat (ITT) principle. ITT analyses on a whole group level will be adjusted for sex, and analyses will also be performed by sex separately. The statistician who performs the ITT analysis will be blinded to group allocation. The number needed to treat will be calculated as the inverted absolute rate reduction for the primary outcomes.

ELIGIBILITY:
Inclusion Criteria for randomized intervention arms A and B:

* Teams participating in youth or adult league series in the 2020 football season. All players in the eligible teams will be invited to participate (players from the age of 14 and older, born 2006 or earlier)
* Teams who have not used a structured training program aiming to prevent injuries that resembles the 3 intervention arms (e.g. the Knee Control program, Knee Control+ program, 11+ program, Adductor strengthening program) on a regular basis the last year
* Teams who have scheduled training at least twice per week

Inclusion criteria for the non-randomized intervention arm C:

* Teams participating in youth or adult league series in the 2020 football season. All players in the eligible teams will be invited to participate (players from the age of 14 and older, born 2006 or earlier)
* Teams who have used the Knee Control program on a regular basis the last year, but no other structured training program aiming to prevent injuries (e.g. the Knee Control+ program, 11+ program, Adductor strengthening program)
* Teams who have scheduled training at least twice per week

Exclusion Criteria:

* Teams who have used a structured groin injury prevention exercise program (e.g. Adductor strengthening program, Hölmich protocol) on a regular basis the last year

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 548 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
All physical complaints injury in four main locations | Study start up to end of season (7 months)
  Any football related injury occurring to the ankle, knee, hamstrings and hip/groin, regardless of need of care or absence from football training or matches ("all physical complaints" injury definition)

SECONDARY OUTCOMES:
All physical complaints injury | Study start up to end of season (7 months)
  Football related injury regardless of need of care or absence from football training or matches ("all physical complaints" injury definition)
Time-loss injury | Study start up to end of season (7 months)
  Football related injury causing absence from training or match with the team ("time-loss injury"). Time-loss injuries will be analyzed for all injury locations and for the four main injury locations (ankle, knee, hamstrings and hip/groin) separately.
Medical attention injury | Study start up to end of season (7 months)
  Football related injury where the player reports seeking care from a medical professional ("medical attention injury"). Medical attention injuries will be analyzed for all injury locations and for the four main injury locations (ankle, knee, hamstrings and hip/groin) separately.
Acute or gradual onset injury | Study start up to end of season (7 months)
  Football related injury that occurs suddenly and is associated with a specific, identifiable event ("acute injury") or injury with gradual onset caused by repeated microtrauma without a single, identifiable event responsible for the injury ("gradual onset injury"). Acute and gradual onset injuries will be analyzed for all injury locations and for the four main injury locations (ankle, knee, hamstrings and hip/groin) separately.
Substantial injury | Study start up to end of season (7 months)
  Football related injury leading to moderate or severe reductions in training volume or performance, or inability to participate in football according to the Oslo Sports Trauma Research Center questionnaire ("substantial injury"). Substantial injuries will be analyzed for all injury locations and for the four main injury locations (ankle, knee, hamstrings and hip/groin) separately.
Adverse events | Study start up to end of season (7 months)
  Adverse events of using the interventions.
Team intervention compliance | Study start up to end of season (7 months)
  Coach reported compliance with each respective intervention protocol. Coaches will report each week the number of team activities (trainings and matches) and the use of the intervention (yes/no) for each of these activities. Team intervention compliance will be calculated as a) the average weekly number of intervention sessions performed during the season, and b) as a proportion, i.e. the number of team intervention sessions / total number of team activities during the season. Team compliance will be reported separately for trainings and matches.
Player intervention compliance | Study start up to end of season (7 months)
  Player reported compliance with each respective intervention protocol. Players will report each week the number of activities (trainings and matches) they participated in and the use of the intervention (yes/no) for each of these activities. Player intervention compliance will be calculated as the average weekly number of intervention sessions performed during the season. Player compliance will be reported separately for trainings and matches.
Exercise fidelity | One observation during the season after approximately 6 months
  Observation of a team training session by a study physiotherapist to evaluate exercise fidelity, i.e. performing exercises according to instructions. A standard checklist will be used in the observation of players performing the intervention exercises and each exercise will be marked as correct/incorrect. Exercise fidelity will be reported as a proportion: number of exercises performed correctly / total number of exercise observations.
Utilization fidelity | Two times during the season: at 4 months and 7 months
  Coach reported utilization fidelity of the intervention. At mid-season (approximately 4 months) and at the end of the season (7 months) coaches will report the use of the intervention program in a survey describing which exercises were used, which progression/difficulty levels of the program were used, timing of the exercise use (before, beginning, during, or after the training session), and dosage (number of sets, number of repetitions or time per exercise). Utilization fidelity will be presented as a descriptive outcome.
Coach experience of injuries and intervention program | Three times during the season: at study start, at 4 months and at 7 months
  Coach baseline, mid-season and follow-up experiences of injuries and of the interventions. Coaches will answer a survey with likert scale questions (rank 1-7) about risk perceptions of sport participation, perceived effects of the intervention, and experiences of using the intervention program. The outcome will be reported as median values of the likert scale questions (1-7).
Player experience of injuries and intervention program | Three times during the season: at study start, at 4 months and at 7 months
  Player baseline, mid-season and follow-up experiences of injuries and of the interventions. Players will answer a survey with likert scale questions (rank 1-7) about risk perceptions of sport participation, perceived effects of the intervention, and experiences of using the intervention program. The outcome will be reported as median values of the likert scale questions (1-7).
Health care need | Study start up to end of season (7 months)
  Number of health care visits due to football related injuries during the season, type of diagnostic examinations and treatments
Costs | Study start up to end of season (7 months)
  Estimated costs of football related injuries and costs of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Martin Hägglund, Professor, Principal Investigator — Linkoeping University
Locations (1):
- Linköping University, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be available upon reasonable request to the principal investigator
Supporting Information: Study Protocol, SAP
Time Frame: Preliminary in autumn 2020
Access Criteria: Study protocol and statistical analysis plan is planned to be submitted in writing to an open access scientific journal

REFERENCES:
- [Derived] Lindblom H, Akerlund I, Walden M, Sonesson S, Hagglund M. Players are positive regarding injury prevention exercise programmes, but coaches need ongoing support: a survey-based evaluation using the Health Action Process Approach model across one season in amateur and youth football. BMJ Open Sport Exerc Med. 2024 Jun 24;10(2):e002009. doi: 10.1136/bmjsem-2024-002009. eCollection 2024. PMID 38933370
- [Derived] Sonesson S, Lindblom H, Hagglund M. Higher age and present injury at the start of the season are risk factors for in-season injury in amateur male and female football players-a prospective cohort study. Knee Surg Sports Traumatol Arthrosc. 2023 Oct;31(10):4618-4630. doi: 10.1007/s00167-023-07517-6. Epub 2023 Aug 5. PMID 37542529
- [Derived] Lindblom H, Walden M, Hagglund M. Adherence to Injury Prevention Exercise Programmes in Amateur Adolescent and Adult Football: A Detailed Description of Programme Use from a Randomised Study. Sports Med Open. 2023 Jul 15;9(1):57. doi: 10.1186/s40798-023-00608-1. PMID 37452894
- [Derived] Lindblom H, Sonesson S, Torvaldsson K, Walden M, Hagglund M. Extended Knee Control programme lowers weekly hamstring, knee and ankle injury prevalence compared with an adductor strength programme or self-selected injury prevention exercises in adolescent and adult amateur football players: a two-armed cluster-randomised trial with an additional comparison arm. Br J Sports Med. 2023 Jan;57(2):83-90. doi: 10.1136/bjsports-2022-105890. Epub 2022 Oct 31. PMID 36316115